CLINICAL TRIAL: NCT04294927
Title: TUBectomy With Delayed Oophorectomy as Alternative for Risk-reducing Salpingo-oophorectomy in High Risk Women to Assess the Safety of Prevention: TUBA-WISP II Study.
Brief Title: TUBectomy With Delayed Oophorectomy in High Risk Women to Assess the Safety of Prevention
Acronym: TUBA-WISP-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Nijmegen (Other)
Responsible Party: Principal Investigator, Joanne A. de Hullu, MD, PhD, Dr. J.A. de Hullu, MD, PhD, University Medical Center Nijmegen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL 70691.091.19
Record Dates: First submitted 2020-03-01; First posted 2020-03-04 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: BRCA1 Gene Mutation; BRCA2 Gene Mutation; RAD51C Gene Mutation; RAD51D Gene Mutation; BRIP1 Gene Mutation; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Risk-reducing salpingectomy with delayed oophorectomy (Experimental): Risk-reducing salpingectomy after the completion of childbearing with delayed oophorectomy.
  Interventions: Procedure: Risk-reducing salpingectomy with delayed oophorectomy
- Risk-reducing salpingo-oophorectomy (Active Comparator): Risk-reducing salpingo-oophorectomy.
  Interventions: Procedure: Risk-reducing salpingo-oophorectomy

INTERVENTIONS:
Procedure: Risk-reducing salpingectomy with delayed oophorectomy — * BRCA1: RRS at age 25-40 and RRO at a maximum age of 45 (advised between 35 and 45).
  * BRCA2: RRS at age 25-45 and RRO at a maximum age of 50 (advised between age 40 and 50).
  * BRIP1, RAD51C, RAD51D: RRS at age 25-50 and RRO at a maximum age of 55 (advised between 45 and 55)
  Arms: Risk-reducing salpingectomy with delayed oophorectomy
Procedure: Risk-reducing salpingo-oophorectomy — * BRCA1 at a maximum age of 40 (advised between age 35 and 40)
  * BRCA2 at a maximum age of 45 (advised between age 40 and 45)
  * BRIP1, RAD51C, RAD51D: at a maximum age of 50 (advised between 45 and 50)
  Arms: Risk-reducing salpingo-oophorectomy

SUMMARY:
The aim of the project is to evaluate the risk-reducing salpingectomy with delayed oophorectomy as an alternative for risk-reducing salpingo-oophorectomy in high risk women with respect to ovarian cancer incidence.

DETAILED DESCRIPTION:
In BRCA1/2 gene mutation carriers, a risk-reducing salpingo-oophorectomy (RRSO) is recommended around the age of 40. This recommendation is based on a 10-40% life-time risk of ovarian cancer in this population and disappointing results of ovarian cancer surveillance for early detection. Moreover, the mortality rate of ovarian cancer is high. Effects of RRSO are a decrease in ovarian cancer risk (80-96%) on one hand and immediate onset of menopause and non-cancer related morbidity on the other hand. The fifty percent breast cancer risk reduction after RRSO has become disputable in the last years. Based on multiple studies showing that most high-grade serous ovarian cancers develop at the distal end of the Fallopian tube, an innovative strategy for RRSO has been developed for this study proposal: risk-reducing salpingectomy (RRS) with delayed risk-reducing oophorectomy (RRO). However, the safety of this strategy has not been proven yet. Before implementing this innovative strategy as standard care we need to investigate the long term effects on ovarian cancer incidence.

ELIGIBILITY:
Inclusion Criteria:

* Women with a class 5 (definitely pathogenic) BRCA1, BRCA2, RAD51C, RAD51D or BRIP1 germline mutation in one of the participating centers.
* Age at inclusion;

  * BRCA1: 25-40 years
  * BRCA2: 25-45 years
  * RAD51C, RAD51D, BRIP1: 25-50 years
* Childbearing completed
* Presence of at least one fallopian tube
* Participants may have a personal history of non-ovarian malignancy
* Informed consent must be obtained and documented according to national and local regulatory requirements and the local rules followed in the institution.

Exclusion Criteria:

* Postmenopausal status (natural menopause or due to treatment)
* Wish for second stage RRO within two years after RRS
* Legally incapable
* Prior bilateral salpingectomy
* A personal history of ovarian, fallopian tube or peritoneal cancer
* Current diagnosis or treatment for malignant disease

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2040-02-17 (Estimated); Study Completion 2040-02-17 (Estimated)

PRIMARY OUTCOMES:
High grade serous (ovarian) cancer incidence | Until the age of 45 for BRCA1 and 50 for BRCA2 germline mutation carriers
  High grade serous (ovarian) cancer incidence

SECONDARY OUTCOMES:
Incidence of (pre)malignant findings in tubes/ovaries | 6 weeks after each surgery
  Incidence of (pre)malignant findings in tubes/ovaries at risk-reducing salpingectomy, oophorectomy and salpingo-oophorectomy.
Peri-operative morbidity and mortality | 6 weeks after each surgery
  Peri-operative morbidity and mortality
Incidence of pelvic cancer (other than ovarian cancer) | Up to the age of 70
  Incidence of pelvic cancer (other than ovarian cancer)
Incidence of breast cancer | Up to the age of 70
  Incidence of breast cancer
Uptake of risk reducing oophorectomy | Up to the age of 70
  Uptake of risk reducing oophorectomy after risk reducing salpingectomy

OTHER OUTCOMES:
High grade serous (ovarian) cancer incidence at the age of 70 | Up to the age of 70
  Exploratory outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Joanne A. de Hullu, MD, PhD, Principal Investigator — Radboud University Medical Center; Karen H. Lu, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center; Rosella P.M.G. Hermens, MD,PhD, Principal Investigator — Radboud University Medical Center; Elizabeth M. Swisher, MD, PhD, Principal Investigator — University of Washington
Locations (48):
- United States (4):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - MD Anderson Cancer Centre, Houston, Texas
  - University of Washington, Seattle, Washington
- Australia (14):
  - Chris O'Brien Lifehouse, Sydney, New South Wales
  - Westmead hospital, Sydney, New South Wales
  - St Andrew War Memorial Hospital, Brisbane, Queensland
  - Royal Brisbane Hospital, Brisbane, Queensland
  - Greenslopes Private Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Frances Perry House, Melbourne, Victoria
  - Mercy Hospital, Melbourne, Victoria
  - Epworth Hospital, Richmon, Victoria
  - Western Health, St Albans, Victoria
  - King Edward Memorial Hospital, Perth, Western Australia
  - Monash Health, Melbourne
  - Peter MacCallum Centre, Melbourne
  - Royal Womens Hospital, Melbourne
- Belgium (2):
  - Hopital Universitaire Bruxelles, Brussels
  - Universitair Ziekenhuis Leuven, Leuven
- AC Camargo Cancer Centre, São Paulo, Brazil
- Italy (3):
  - Universita di Bologna, Bologna
  - San Gerardo Hospital, Monza
  - Gemelli Hospital, Rome
- Instituto Nacional de Cancerología, Mexico City, Mexico
- Netherlands (14):
  - Radboudumc, Nijmegen, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg, North Brabant
  - Amsterdam University Medical Center, Amsterdam
  - Antoni van Leeuwenhoek, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Medical Center Leeuwarden, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht
  - Maxima Medical Center, Veldhoven
  - Isala Klinieken, Zwolle
- Norway (3):
  - Akershus University Hospital, Nordbyhagen
  - Oslo University Hospital, Oslo
  - Stavanger Uniersity Hospital, Stavanger
- Poland (4):
  - Gdynia Oncology Centre, Gdynia
  - Bonifraterskie Centrum Medyczne, Katowice
  - Medical University of Silesia, Katowice
  - National Cancer Institute Warsaw, Warsaw
- Karolinksa Institutet, Stockholm, Sweden
- Hospital Británico, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pennington KP, Pugh SL, Huh W, Walker JL, Jewell E, Havrilesky LJ, Carter J, Muller CY, Drapkin R, Lankes HA, Castellano T, Zamorano AS, Blank SV, Kachnic LA. Optimization of Timing for Risk-Reducing Salpingectomy and Oophorectomy. Obstet Gynecol. 2025 Jan 1;145(1):21-30. doi: 10.1097/AOG.0000000000005781. Epub 2024 Nov 7. PMID 39509704
- [Derived] Steenbeek MP, van Bommel MHD, intHout J, Peterson CB, Simons M, Roes KCB, Kets M, Norquist BM, Swisher EM, Hermens RPMG; TUBA-WISP II consortium; Lu KH, de Hullu JA. TUBectomy with delayed oophorectomy as an alternative to risk-reducing salpingo-oophorectomy in high-risk women to assess the safety of prevention: the TUBA-WISP II study protocol. Int J Gynecol Cancer. 2023 Jun 5;33(6):982-987. doi: 10.1136/ijgc-2023-004377. PMID 37045546